CLINICAL TRIAL: NCT06358781
Title: Screening Whole Grain Dietary Intake Biomarkers and Validating the Dose-response Relationship in a Randomized Controlled Study in China.
Brief Title: A Dose-response Study to Validate the Biomarkers for Whole Grain Dietary Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: xuyajun197673-002
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Chronic Disease Prevention
Keywords: Whole grain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (WG wheat flour intake= 0 g) (No Intervention): An acute randomized controlled trial was performed and the total study group is randomly divided into four groups: the amounts of WG wheat flour for group A were 0 g.
- Group B (WG wheat flour intake= 25 g) (Experimental): An acute randomized controlled trial was performed and the total study group is randomly divided into four groups: the amounts of WG wheat flour for group B were 25 g.
  Interventions: Other: Whole grain wheat flour
- Group C (WG wheat flour intake= 50 g) (Experimental): An acute randomized controlled trial was performed and the total study group is randomly divided into four groups: the amounts of WG wheat flour for group C were 50 g.
  Interventions: Other: Whole grain wheat flour
- Group D (WG wheat flour intake= 100 g) (Experimental): An acute randomized controlled trial was performed and the total study group is randomly divided into four groups: the amounts of WG wheat flour for group D were 100 g.
  Interventions: Other: Whole grain wheat flour

INTERVENTIONS:
Other: Whole grain wheat flour — Group A: whole grain flour: 0 g Group B: Whole grain flour: 25 g Group C: Whole grain flour: 50 g Group D: whole grain flour: 100g
  Arms: Group B (WG wheat flour intake= 25 g); Group C (WG wheat flour intake= 50 g); Group D (WG wheat flour intake= 100 g)

SUMMARY:
Dose-response validation of whole grain dietary intake biomarkers remains limited, and it is debatable whether these markers could be utilized as classifiers for different levels of whole grain consumption. Because there are significant disparities in genetic background and dietary patterns between Chinese and Western cultures, it is unclear if whole grain dietary intake biomarkers can characterize whole grain consumption in Chinese populations. To address these issues, the current study was designed to evaluate the sensitivity and specificity of potential whole grain markers in a randomized controlled trial, as well as to validate the markers' dose-response relationship, so that they can be used in nutritional epidemiological studies and dietary intake assessments of whole grains.

DETAILED DESCRIPTION:
An acute randomized controlled trial was performed and the total study group is randomly divided into four groups: the amounts of WG wheat flour administered were 0 g, 25g, 50 g and 100 g. Experimental period with a total of 6 days was subdivided into two parts: -5 days to 0 h defined as the run-in period, 0-24 h (after the dose-related test meal), defined as the test day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* age 18-40 years
* BMI 18.5-23.9 kg/m2.

Exclusion Criteria:

* pregnancy or breastfeeding
* vegetarian;
* smokers;
* acute and chronic diseases;
* allergic to wheat;
* frequent nutrients supplement use;
* medication use of antibiotics within 1-month;
* more than 3 kg weight change within 3-month;
* unwillingness to follow dietary restrictions;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
whole grain plasma and urine biomarkers discovery and identification | Baseline and 0~24 hours after intervention food intake
  Discovery of whole grain plasma and urine biomarkers after acute intakes of WG wheat food using LC-MS untargeted metabolomics approach in a designed study, identify the specific biomarkers for WG wheat with high confidence levels.

SECONDARY OUTCOMES:
Validate the performance of the potential WG biomarkers. | Baseline and 0~24 hours after intervention food intake
  The receiver operating characteristic analysis was used to validate the performance of the potential WG biomarkers in the dose-response validation set

OTHER OUTCOMES:
Dose-response of WG wheat biomarkers. | Baseline and 0~24 hours after intervention food intake
  Linear regression analysis was performed between WGs amount consumed and the average concentration for each WG biomarkers, giving a regression equation and r2 values.

CONTACTS AND LOCATIONS:
Overall Officials: Yajun Xu, Study Director — Peking University
Locations (1):
- Department of Nutrition and Food Hygiene, School of Public Health, Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Shared results in a publication
Supporting Information: Study Protocol
Time Frame: Expected after publication (December 2024)
Access Criteria: In a publication